CLINICAL TRIAL: NCT06134895
Title: Randomised Double Blind Comparison of Prophylactic Tramadol and Tramadol Plus Ketamine for Prevention of Shivering After Spinal Anesthesia in Lower Segment Caeserian Section
Brief Title: Tramadol and Tramadol Plus Ketamine for Shivering Prevention After Spinal Anesthesia in Lower Segment Caeserian Section
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ziauddin University (Other)
Responsible Party: Principal Investigator, Dr Muhammad Arif, Principal Investigator, Ziauddin University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 7240623MAANE
Record Dates: First submitted 2023-09-11; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-11

CONDITIONS: Shivering
Keywords: Shivering; Anesthesia, Spinal; Caesarean
MeSH Terms: interventions — Tramadol; Ketamine

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tramadol with Ketamine (Experimental): Tramadol 0.25mg/Kg with Ketamine 0.25 mg/Kg
  Interventions: Drug: Tramadol with Ketamine
- Tramadol (Active Comparator): Tramadol 0.5mg/kg
  Interventions: Drug: Tramadol

INTERVENTIONS:
Drug: Tramadol with Ketamine — Tramadol with Ketamine is being provided randomly using prospective, double-blind
  Arms: Tramadol with Ketamine
Drug: Tramadol — Tramadol alone is being provided randomly using prospective, double-blind
  Arms: Tramadol

SUMMARY:
The objective of this study is to compare the efficacy of prophylactic use of intravenous tramadol versus tramadol plus ketamine for prevention of shivering under spinal anaesthesia in lower segment caeserian section.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 40 years
* American Society of Anesthesiologist physical status I and II
* Pregnant female for lower segment caeserian section

Exclusion Criteria:

* Patients with Hypertension
* Patients with hypo- or hyperthyroidism
* Known case of Cardiopulmonary disease, pre-eclampsia and eclampsia
* An initial body temperature 38.00C or, 36.0oC assessed by thermometer

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 190 (Estimated)
Dates: Start 2023-08-16 (Actual); Primary Completion 2023-11-16 (Estimated); Study Completion 2023-11-16 (Estimated)

PRIMARY OUTCOMES:
Incidence of shivering | Patients will be monitored from 15-45 mins from the administration of the prophylactic drug
  Muscular activity in one or more than one muscle group or involving the whole body will be labelled as shivering
Severity of Shivering | Patients will be monitored from 15-45 mins from the administration of the prophylactic drug
  Shivering will be graded as per the following criteria:
  0= no shivering.
  1. piloerection or peripheral vasoconstriction but no visible shivering.
  2. muscular activity (visible muscular twitching) in only one muscle group;
  3. muscular (visible muscular twitching) activity in more than one muscle group but not generalized.
  4. shivering involving the whole body

SECONDARY OUTCOMES:
Time to shivering | 15 mins from the administration of the prophylactic drug
  The time to shiver will be defined as the duration from the initiation of the intervention until the onset of observable shivering.
Complications | Patients will be monitored from 15-45 mins from the administration of the prophylactic drug
  Complications such as hypotension, nausea and vomiting, bradycardia, or hallucinations will be noted

CONTACTS AND LOCATIONS:
Overall Officials: Muhammad Arif, Principal Investigator — Ziauddin University
Locations (1):
- Muhammad Arif, Karachi, Sindh, Pakistan

IPD SHARING:
Plan to Share IPD: No